CLINICAL TRIAL: NCT05773638
Title: Cardiovascular and Venous Thromboembolism Disease in Patients with Von Willebrand Disease in the French West
Acronym: TWIGO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TWIGO ( 29BRC21.0204)
Record Dates: First submitted 2023-02-21; First posted 2023-03-17 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Von Willebrand Diseases
Keywords: von Willebrand disease; venous thromboembolism disease; cardiovascular disease; atrial fibrillation
MeSH Terms: conditions — von Willebrand Diseases; Cardiovascular Diseases; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Due to increasing of life expectancy, patients with von Willebrand disease are exposed to age-related pathologies such as cancer or cardiovascular diseases. Management of thrombotic events is challenging given the inherent bleeding risk in von Willebrand disease. Few data are currently available in the literature.

The aim of the study is to describe the frequency and nature of arterial and venous thromboembolic events and atrial fibrillation in patients with von Willebrand disease in the West of France.

The investigators will perform a retrospective multicenter study conducted in the von Willebrand population of the French West. Von Willebrand adult patients followed in one of the French West medical centers participating in the study, who presented deep vein thrombosis, pulmonary embolism, ischemic stroke, transient ischemic attack, acute coronary syndrome, acute limb ischemia, atrial fibrillation, arteriopathy of the lower limbs, angina will be eligible.

DETAILED DESCRIPTION:
Von Willebrand disease is the most common hereditary bleeding disorder. Due to the development of therapies, life expectancy and life quality are increasing in affected patients. However, certain treatments and/or certain comorbidities associated with venous and arterial thrombotic risks may be present in these patients. In the general population, venous thromboembolic disease, arterial thrombosis and atrial fibrillation are frequent. Their management requires the use of antiaggregants and anticoagulant molecules, themselves associated with a bleeding risk. Few data are currently available in the literature concerning the occurrence of venous and arterial thromboembolic events in patients with von Willebrand disease and their management, in the face of a hemorrhagic risk inherent to their pathology and its increase by anti-aggregant treatments and anticoagulants.

The aim of the study is to describe the frequency and nature of arterial and venous thromboembolic events and atrial fibrillation in patients with von Willebrand disease in the West of France.

The investigators will perform a retrospective multicenter study on data conducted in the French West. The study population is composed of patients with von Willebrand disease followed in a reference center in the French West, have consented to be included in the BERHLINGO database (Base d'Etude et de Recherche pour Les INvestigateurs en Hémostase du Grand-Ouest), and who presented deep vein thrombosis, pulmonary embolism, ischemic stroke, transient ischemic attack, acute coronary syndrome, acute limb ischemia, atrial fibrillation, arteriopathy of the lower limbs, angina. Data about von Willebrand disease, risk factors, event, treatment such as antiaggregants and anticoagulants and complications such as hemorrhage or recurrence, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Von Willebrand disease
* Adult
* Followed-up in a reference center of West of France (Caen, Brest, Nantes, Rennes, Le Mans, Angers)
* Consented to be included in BERHLINGO database
* Have presented a thrombotic and/or embolic event or cardiovascular disease including deep vein thrombosis, pulmonary embolism, ischemic stroke, transient ischemic attack, acute coronary syndrome, acute limb ischemia or angina or obliterating arteriopathy of the lower limbs, atrial fibrillation.
* Have not expressed their opposition

Exclusion Criteria:

* - Expression of opposition
* Acquired von Willebrand syndrome
* Patients under legal protection
* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with von Willebrand disease followed in a reference center in the French West and who have consented to be included in the BERHLINGO database (Base d'Etude et de Recherche pour Les INvestigateurs en Hémostase du Grand-Ouest) with a medical history of deep vein thrombosis, pulmonary embolism, ischemic stroke, transient ischemic attack, acute coronary syndrome, acute limb ischemia, angina, obliterating arteriopathy of the lower limbs or atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-26 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
To describe the frequency of arterial and venous thromboembolic events and cardiac arrhythmia due to atrial fibrillation in patients with Willebrand disease in the Greater West. | 12 months
  Occurrence of a thromboembolic event validated by an adjudication committee
To describe the nature of arterial and venous thromboembolic events and cardiac arrhythmia due to atrial fibrillation in patients with Willebrand disease in the Greater West. | 12 months
  Occurrence of a thromboembolic event validated by an adjudication committee

SECONDARY OUTCOMES:
Identify potential risk factors | 12 months
  identify whether certain risk factors are more prevalent in the population than others
Number of revascularisation procedures, anticoagulants and antiaggregants prescribed for these conditions | 12 months
  Prescription of anticoagulant and/or antiaggregant treatment
Evaluate the nature of treatments prescribed for these pathologies: revascularisation procedures, anticoagulants and antiaggregants | 12 months
  Revascularisation procedure (endovascular or surgical)
Evaluate the tolerance of these treatments | 12 months
  Occurrence of clinical haemorrhage
Evaluate the effectiveness of these treatments | 12 months
  Occurrence of a cardio-embolic event
Evaluate the effectiveness of these treatments | 12 months
  Occurrence of a thromboembolic recurrence
Evaluate the effectiveness of these treatments | 12 months
  Death from haemorrhage and/or thromboembolic causes.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CH le MANS, Le Mans
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three month and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.